CLINICAL TRIAL: NCT01552538
Title: Long Term Observational Study of the Safety and Efficacy of an Active Implantable Vagal Nerve Stimulation Device in Patients With Rheumatoid Arthritis
Brief Title: Long Term Extension Study For SPM-005 Participants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPM-006
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Vagus Nerve; Vagal Nerve Stimulation
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyberonics VNS System (Experimental): Continued stimulation w/Cyberonics VNS
  Interventions: Device: Cyberonics VNS System

INTERVENTIONS:
Device: Cyberonics VNS System — Stimulation with an active implantable electrical vagal nerve stimulation device

SUMMARY:
This will be an open label multicenter study of the safety and efficacy of an active implantable vagal nerve stimulation (VNS) device in patients with rheumatoid arthritis. Patients who complete study SPM-005 will be enrolled in this study at the time of the last visit of the preceding study.

DETAILED DESCRIPTION:
This will be an open label multicenter study of the safety and efficacy of an active implantable vagal nerve stimulation (VNS) device in patients with rheumatoid arthritis.

Patients who complete study SPM-005 will be enrolled in this study at the time of the last visit of the preceding study. The assessments at the last visit of the preceding study will also be used as baseline measures for the current study. If the patient has previously discontinued SPM-005 and greater than 30 days have elapsed since the final visit in SPM-005, baseline measures for the current study will be repeated, and an interim medical history will be taken to assess whether any new medical conditions were diagnosed in the time between studies.

Follow-up visits will occur at 3, 6, 12, 18, 24, 36 and 48 months. A final follow-up visit will occur for all remaining patients at study closure when the final enrolled subject has completed 48 months on study.

The study will continue until the last patient entered has completed 48 months in this study.

An Interim Visit or a phone contact must be performed a maximum of 2 months after any change in device settings. Interim visits may also be performed at any time at the investigator's discretion; either between scheduled visits, or after the patient has completed the Month 48 Visit, if the study is still ongoing.

The primary efficacy objective is to determine the long term efficacy of vagal nerve stimulation as assessed by the DAS28 score.

The secondary efficacy objectives are to determine the long term efficacy of vagal nerve stimulation as assessed by:

* the ACR 20, 50 and 70 response rate,
* the EULAR response rate, and
* changes in the Euro-QoL score.

The safety objectives are to determine the long term safely of vagal nerve stimulation as assessed by the subject incidence rates of:

* Adverse events
* Serious adverse events
* Device deficiencies

ELIGIBILITY:
Inclusion Criteria:

* Patients must have participated in study SPM-005

Exclusion Criteria:

* Inability to provide informed consent
* Significant psychiatric illness or substance abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-05 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Change in rheumatoid arthritis Disease Activity Score (DAS) from baseline visit | 12-18 months

SECONDARY OUTCOMES:
Subject incidence of Adverse Events | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Zitnik, M.D., Study Director — SetPoint Medical
Locations (4):
- Bosnia and Herzegovina (2):
  - Sveučilišna klinička bolnica Mostar, Mostar
  - Klinicki Centar Univerziteta, Reumatologija, Sarajevo
- Sisters of Mercy Clinical Hospital Centre, Zagreb, Croatia
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No